CLINICAL TRIAL: NCT06212986
Title: Enhancing Psychological Skills and Well-being in Sport Through a Blended Intervention: a Controlled Study With Perform-UP Tennis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Daniela Villani, Associate Professor of General Psychology, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 4221_2021
Record Dates: First submitted 2023-12-23; First posted 2024-01-19 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Psychological Well-Being
Keywords: mobile app; psychological well-being; sport; tennis players
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental blended group (Experimental): The experimental blended group (perform-up group) used the application Perform-UP Tennis on their own and also met up with a professional sports psychologist every 2 weeks for debriefing. Participants were asked to answer a series of questionnaires in two separate phases.
  Interventions: Device: Promotion of mental training through mobile application Perform-UP Tennis
- Control group (No Intervention): Participants were asked to answer a series of questionnaires in two separate phases, but they only carried out their classic technical training without integrating the mental training program with the app Perform-UP Tennis.

INTERVENTIONS:
Device: Promotion of mental training through mobile application Perform-UP Tennis — Perform-UP Tennis is a sport specific mental training app that integrates breathing, relaxation and na-ture-based guided imagery exercises and aims to promote emotional well-being and the enhancement of mental skills. The app techniques are integrated into a single gradual path that involves increasingly complex breathing and relaxation exercises with increasing duration.
  The intervention consists of eight weekly modules over a period of 8 weeks with progressive exercises.
  Arms: Experimental blended group

SUMMARY:
Mental preparation is a fundamental aspect of athletic performance. The investigators present here an experiment aimed at evaluating the effectiveness of a blended intervention to promote mindfulness and self-confidence and a reduction of anxiety among professional athletes. Perform-UP Tennis is an application that provides a weekly mental training program to be integrated into the athlete's daily routine. The intervention included eight weekly modules with variable and progressive training and relaxation exercises. Meetings with the athletes took place every 2 weeks. The study involved 41 tennis players who were randomly assigned to either the intervention or the control group.

ELIGIBILITY:
Inclusion Criteria:

* being tennis players with a minimum age of 14
* being fluent in Italian
* having a smartphone with an Internet connection

Exclusion Criteria:

* having hearing difficulties
* not playing tennis
* being younger than 14 years old
* not having a good knowledge of Italian

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
The Psychological Inventory of Sport Performance (IPPS-48) was used to assess athletes' mental abilities. The questionnaire included 48 items, divided into eight subscales each reflecting eight mental abilities. | It was assessed at baseline (T0) and after eight weeks, which is at the end of the intervention (T1)
  Each scale included five items, to which the athletes responded on a 5-point Likert scale. The eight subscales reflected the following eight mental abilities: concentration, arousal control, preparation of the match, goal setting, visualization, cognitive anxiety, self-confidence and self-talk. But for this research, the investigators considered only three subscales that were consistent with the activities proposed within the application (breathing and relaxation techniques). The scales considered were: cognitive anxiety, which evaluates the athlete's level of concern during the match, fear of making mistakes, and fear of failing, self-confidence, which evaluates the confidence that the athlete has in being able to compete at his/her best, to give their best and to believe in themselves, emotional arousal control, which evaluates the athlete's ability to relax when he/she feels anxious and under tension and to activate him/herself when he/she needs to reach the right energy level.
The Mindfulness Inventory for Sport (MIS) was used to evaluate the awareness processes within the athlete's sports performance. The scale consists of 15 items reflecting three distinct components of mindfulness. | It was assessed at baseline (T0) and after eight weeks, which is at the end of the intervention (T1)
  Each scale included five items, to which the athletes responded on a 5-point Likert scale. It contains both positively and negatively worded items (the non-judgmental subscale was reverse-scored). Specifically, this questionnaire assessed: (1) Awareness, being aware of stimuli and their associated internal reactions, (2) non-judgmental, adopting a non-judgmental attitude towards these stimuli and reactions, (3) refocusing, quickly refocus attention on target signals.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Sacred Heart, Milan, Italy

REFERENCES:
- [Derived] Bordo S, Costanzo G, Villani D. Enhancing psychological skills and well-being in sport through an app-based blended intervention: a randomized controlled pilot study. BMC Psychol. 2025 May 21;13(1):537. doi: 10.1186/s40359-025-02824-8. PMID 40400025